CLINICAL TRIAL: NCT06211855
Title: Cerebroplacental Ratio and Perinatal Outcomes in Mild and Moderate Idiopathic Polyhydramios Cases
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, şükran doğru, medical doctor, fellowship, Necmettin Erbakan University
Other Study IDs: 2023/4702 (17181
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Idiopathic Polyhydramios Cases
Keywords: polyhidramnios,cerebroplacental ratio

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic Polyhydramios Cases: The group with polyhydramnios was divided into two groups according to whether the CPR value was below 1.08 or 1.08 and above
  Interventions: Diagnostic Test: doppler assesment
- low-risk pregnant women: The control group included low-risk pregnant women who did not have polyhydramnios. Women who had chromosomal or anatomical abnormalities, multiple pregnancies, oligohydramnios (AFI 5 cm), severe polyhydramnios, fetal growth restriction, elective cesarean section (CS), pre-existing conditions (hypertension, diabetes, thrombophilia), or obstetric complications (gestational hypertension, preeclampsia, gestational diabetes) were excluded.
  Interventions: Diagnostic Test: doppler assesment

INTERVENTIONS:
Diagnostic Test: doppler assesment — In all cases, the measurement, including UA PI and MCA PI, was measured with a 6-4 MHz convex transabdominal probe. All measurements were made by an obstetrician (Ş.D.) with 28 years of experience. Doppler measurements were collected from the proximal third of the MCA and the free-floating segment of the umbilical cord, ensuring that the angle of insonation was as close to zero as feasible and that fetal movements were absent

SUMMARY:
This study aims to evaluate the predictability of fetal Doppler parameters in terms of perinatal adverse outcomes in singleton pregnancies with mild and moderate idiopathic polyhydramnios

DETAILED DESCRIPTION:
Pregnant women diagnosed with mild-moderate IP and randomly selected low-risk singleton pregnancies without polyhydramnios were included in the study one-on-one by matching their gestational ages. The diagnosis of polyhydramnios was made if the AFI was 24 cm and above.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with mild-moderate IP ,selected low-risk singleton pregnancies without polyhydramnios

Exclusion Criteria:

* Women who had chromosomal or anatomical abnormalities, multiple pregnancies, oligohydramnios (AFI 5 cm), severe polyhydramnios, fetal growth restriction, elective cesarean section (CS), pre-existing conditions (hypertension, diabetes, thrombophilia), or obstetric complications (gestational hypertension, preeclampsia, gestational diabetes) were excluded

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women diagnosed with mild-moderate IP and randomly selected low-risk singleton pregnancies without polyhydramnios were included in the study one-on-one by matching their gestational ages.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
perinatal outcome | 1 year
  adverse perinatal outcome: The week of birth and type of birth of all pregnant women participating in the study will be recorded. Premature birth rates and reasons for cesarean section will be questioned in all pregnant women. Birth weights of all neonates, 1st and 5th minute Apgar scores, and admissions to the neonatal intensive care unit will be recorded. Necessary statistical evaluation will be made in all healthy and polyhydramnios cases.

CONTACTS AND LOCATIONS:
Overall Officials: şükran doğru, Principal Investigator — NECMETTİN ERBAKAN UNIVERCITY
Locations (1):
- Necmettin Erbakan University, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
shared when the work is completed
Supporting Information: Study Protocol
Time Frame: 01-01-2023 30-11-2023
Access Criteria: ıd